CLINICAL TRIAL: NCT06836349
Title: Registry-randomized Comparison of Rehabilitation Regimens After Flexor Pollicis Longus Injury in the Thumb
Brief Title: Registry-randomized Comparison of Rehabilitation Regimens After Flexor Tendon Injury in the Thumb
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Region Östergötland (Other); Region Västerbotten (Other Government); Region Örebro County (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Maria Wilcke, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRCT HAKIR fpl
Record Dates: First submitted 2025-02-07; First posted 2025-02-20 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Flexor Tendon Injury; Rehabilitation Program; Flexor Tendon Rupture; Thumb Injury
Keywords: Flexor pollicis longus injury; RRCT; Early active motion; flexor tendon injury; Thumb; Immobilisation
MeSH Terms: interventions — Immobilization; Casts, Surgical

STUDY DESIGN:
Intervention Model Description: Registry-randomized controlled trial (RRCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early active motion (Active Comparator): Early active motion 2-5 days postoperatively.
  Interventions: Other: Early active motion training after operated FPL injury
- Immobilisation in plaster cast 4 weeks (Active Comparator): Immobilisation in plaster cast 4 weeks postoperatively
  Interventions: Other: Immobilisation in plaster cast 4 weeks after operated FPL injury

INTERVENTIONS:
Other: Early active motion training after operated FPL injury — Early active motion training after operated FPL injury
  Arms: Early active motion
Other: Immobilisation in plaster cast 4 weeks after operated FPL injury — Immobilisation in plaster cast 4 weeks after operated FPL injury
  Arms: Immobilisation in plaster cast 4 weeks

SUMMARY:
Flexor tendon injuries in the thumb occur across all ages and genders. Each year, approximately 400 patients undergo surgery for a flexor tendon injury in Sweden. These injuries are exclusively treated at one of the seven specialized hand surgery clinics, as the surgery is technically demanding, and postoperative rehabilitation is critical, specialized, and requires expertise from hand therapists. To prevent tendon adhesions and stiffness in the thumb or fingers, controlled active motion therapy is usually initiated within a few days after surgery. Studies on finger flexor tendon injuries have shown that early active movement therapy leads to better mobility compared to immobilization. Consequently, early active training is now the standard treatment following flexor tendon repair. However, during postoperative rehabilitation, the repaired flexor tendon may rupture, often necessitating revision surgery.

The rupture rate after flexor tendon repair in the thumb is approximately three times higher than in other fingers (10% vs. 3%). While most studies on flexor tendon injuries focus on finger tendons, research on the outcomes of thumb flexor tendon injuries is limited. The biomechanics and anatomy of the thumb's flexor tendon differ significantly from those of finger tendons.

The objective of this study is to determine whether the rupture rate following thumb flexor tendon surgery can be reduced by immobilizing the thumb in a cast for four weeks postoperatively, compared to standard early active motion therapy, without negatively affecting joint mobility and thumb strength. Additionally, the study will evaluate patient-reported outcomes one year post-surgery for both rehabilitation regimens (immobilization vs. mobilization).

This study is a registry-randomized clinical trial (RRCT) involving five hand surgery clinics in Sweden. Data following randomization between the two rehabilitation protocols will be collected through follow-up in the Swedish National Hand Surgery Quality Registry (HAKIR).

ELIGIBILITY:
Inclusion Criteria:

Complete laceration of the thumb flexor tendon (Flexor Pollicis Longus; FPL) within zone 1 and 2.

Age over 15 years. Minors (<18 years) are considered to have sufficient maturity to understand the implications of the research.

Swedish-speaking / able to understand spoken and written Swedish. Surgery performed within 14 days from the time of injury.

Exclusion Criteria:

Tendon injury with a defect requiring tendon grafting. Another complete tendon injury in the same hand. Extensive associated injuries, such as fracture, vascular injury with circulatory impairment, large skin defect, or preoperative signs of infection. Patient deemed unsuitable for early active motion therapy due to factors such as lack of cooperation, cognitive impairment, or substance abuse issues.

Patient declines follow-up in the HAKIR quality registry. Wound infection making early active motion therapy inappropriate.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Tendon rupture rate | Within one year after operation
  Clinically diagnosed rupture of an operated flexor pollicis longus injury

SECONDARY OUTCOMES:
Active range of motion in the joints of the operated thumb MCP joint | 3 and 12 months postoperatively
  Active range of motion of the MCP joint of the operated thumb measured with a goniometer
Active range of motion of the IP-joint in the opererated thumb | 3 and 12 months postoperatively
  Measured with a goniometer
Grip strength | 3 and 12 months postoperatively
  Measured using a Jamar dynamometer and compared to the uninjured side.gauge.
Key pinch strength | 3 and 12 months postoperatively
  Key pinch between the thumb and index finger assessed with a pinch gauge.
HQ-8 questionnaire | 3 and 12 months postoperatively
  A Patient-rated outcpme measurs (PROM).The HAKIR questionnaire (HQ-8) consists of seven questions regarding symptoms in the operated hand, such as aching, pain, numbness, weakness, and cold sensitivity, as well as one question on perceived hand function. All questions are answered on a 0-100 scale (0, 10, 20, etc.). An additional question in the questionnaire addresses satisfaction with the surgical outcome and the experience of staff interactions during the given care, rated from completely dissatisfied to completely satisfied.
Quick DASH | 3 and 12 months postoperatively
  A patient-rated outcpme measure. (PROM. The short version of the Disabilities of the Arm, Shoulder, and Hand (QuickDASH) contains 11 questions covering activity limitations, symptoms, and participation. The responses are summed into a total score ranging from 0 to 100, where 100 represents maximum perceived disability of the hand and arm.

CONTACTS AND LOCATIONS:
Locations (5):
- Sweden (5):
  - Hand- och plastikkirurgiska kliniken Linköpings Universitetssjukhus, Linköping
  - Handkirurgiska kliniken Örebros Universitetssjukhus, Örebro
  - Handkirurgiska kliniken Södersjukhuset, Stockholm
  - Handkirurgiska kliniken Norrlands Universitetssjukhus, Umeå
  - Handkirugiska kliniken Uppsala Akademiska Sjukhus, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data might be shared upon request for metaanalyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the results are analyzed and publish and 10 years ahead
Access Criteria: Researchers with an ethical permitt, as descibed above, by request to maria.wilcke@ki.se